CLINICAL TRIAL: NCT02601612
Title: A Phase I Study of the Safety and Immunogenicity of a Single Dose of the Live Recombinant RSV D46cpΔM2-2 Vero Grown Virus Vaccine (Lot RSV #008A), Delivered as Nose Drops to RSV-Seropositive Children 12 to 59 Months of Age and RSV-Seronegative Infants and Children 6 to 24 Months of Age
Brief Title: Safety and Immunogenicity of the RSV D46cpΔM2-2 Vaccine in RSV-Seropositive Children and RSV-Seronegative Infants and Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR 308
Record Dates: First submitted 2015-11-09; First posted 2015-11-10 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1: D46cpΔM2-2 Vaccine (Experimental): RSV-seropositive children will receive a single dose of 10^6 PFU D46cpΔM2-2 vaccine at study entry (day 0).
  Interventions: Biological: D46cpΔM2-2 vaccine
- Group 1: Placebo (Placebo Comparator): RSV-seropositive children will receive a single dose of placebo at study entry (day 0).
  Interventions: Biological: Placebo
- Group 2: D46cpΔM2-2 Vaccine (Experimental): RSV-seronegative infants and children will receive a single dose of 10^5 PFU D46cpΔM2-2 vaccine at study entry (day 0).
  Interventions: Biological: D46cpΔM2-2 vaccine
- Group 2: Placebo (Placebo Comparator): RSV-seronegative infants and children will receive a single dose of placebo at study entry (day 0).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: D46cpΔM2-2 vaccine — Delivered as nose drops
  Arms: Group 1: D46cpΔM2-2 Vaccine; Group 2: D46cpΔM2-2 Vaccine
Biological: Placebo — Delivered as nose drops
  Arms: Group 1: Placebo; Group 2: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of the RSV D46cpΔM2-2 vaccine in RSV-seropositive children and RSV-seronegative infants and children.

DETAILED DESCRIPTION:
Human RSV is the most common viral cause of serious acute lower respiratory illness (LRI) in infants and children under 5 years of age worldwide. This study will evaluate the safety and immunogenicity of the RSV D46cpΔM2-2 vaccine in RSV-seropositive children and RSV-seronegative infants and children. The vaccine will be evaluated in a stepwise fashion beginning in RSV-seropositive children (Group 1), and then in RSV-seronegative infants and children (Group 2). In each group, participants will be randomly assigned to receive a single dose of D46cpΔM2-2 vaccine or placebo at study entry (day 0).

Participants will be enrolled in the study between April 1 and October 31, outside of the RSV season. Group 1 (RSV-seropositive children) will attend several study visits and will be followed for 28 days. Group 2 (RSV-seronegative infants and children) will remain on study until they complete the post-RSV season visit between April 1 and April 30 in the calendar year following enrollment. Participants in Group 2 will also attend several study visits during the time they are enrolled in the study. Study visits for all participants may include clinical assessments, blood collection, and nasal washes.

ELIGIBILITY:
RSV-Seropositive Children:

Inclusion Criteria:

* Greater than or equal to 12 months of age and less than 60 months of age
* Received routine immunizations appropriate for age
* Serum RSV neutralizing antibody titer greater than or equal to 1:40
* Serum RSV neutralizing antibody result obtained this calendar year
* Pre-inoculation serum RSV neutralizing antibody specimen obtained less than or equal to 56 days prior to inoculation
* Parent/guardian has completed the study comprehension assessment
* Parent/guardian has signed the study informed consent document (ICD)
* Subject is expected to be available for the duration of the study

Exclusion Criteria:

* Evidence of chronic disease
* Within the past 6 months had a decline in height or weight growth that crosses two major growth percentiles (e.g., from above the 75th to below the 25th)
* Known or suspected impairment of immune function
* Maternal history of positive HIV test
* Bone marrow/solid organ transplant recipient
* Major congenital malformations, including congenital cleft palate or cytogenetic abnormalities
* Current or unresolved suspected or documented developmental disorder, delay, or other developmental problem
* Cardiac abnormality requiring treatment
* Lung disease or reactive airway disease
* More than one episode of wheezing in the first year of life
* Wheezing episode or received bronchodilator therapy within the past 12 months
* Previous immunization with an experimental RSV vaccine
* Previous receipt or planned administration of anti-RSV antibody product
* Previous serious vaccine-associated AE or anaphylactic reaction
* Known hypersensitivity to any vaccine component
* Previous receipt of immunoglobulin or any antibody products
* Previous receipt of any other blood products within the past 6 months
* Member of a household that contains an infant who is less than 12 months of age during study days 0 to 10
* Member of a household that includes an immunocompromised individual
* Member of a household that includes a person who has received chemotherapy within the past 12 months
* Will attend a daycare facility that does not separate children by age and contains an infant who is greater than 12 months of age during study days 0 to 10

RSV-Seronegative Infants and Children:

Inclusion Criteria:

* Greater than or equal to 6 months of age and less than 25 months of age
* Received routine immunizations appropriate for age
* Serum RSV neutralizing antibody titer is less than 1:40
* Screening and pre-inoculation serum RSV neutralizing antibody specimen obtained less than or equal to 42 days prior to inoculation
* Parent/guardian has completed the study comprehension assessment
* Parent/guardian has signed the study ICD
* Subject is expected to be available for the duration of the study
* Born at greater than or equal to 37 weeks gestation or is currently greater than 1 year of age

Exclusion Criteria:

* Evidence of chronic disease
* Within the past 6 months had a decline in height or weight growth that crosses two major growth percentiles (e.g., from above the 75th to below the 25th)
* Known or suspected impairment of immune function
* Maternal history of positive HIV test
* Bone marrow/solid organ transplant recipient
* Major congenital malformations, including congenital cleft palate or cytogenetic abnormalities
* Current or unresolved suspected or documented developmental disorder, delay, or other developmental problem
* Cardiac abnormality requiring treatment
* Lung disease or reactive airway disease
* More than one episode of wheezing in the first year of life
* Wheezing episode or received bronchodilator therapy within the past 12 months
* Previous immunization with an experimental RSV vaccine
* Previous receipt or planned administration of anti-RSV antibody product
* Previous receipt of immunoglobulin or any antibody products
* Previous receipt of any other blood products within the past 6 months
* Previous serious vaccine-associated AE or anaphylactic reaction
* Known hypersensitivity to any vaccine component
* Member of a household which contains an infant who is less than 6 months of age during study days 0 to 28
* Member of a household that includes an immunocompromised individual
* Member of a household that includes a person who has received chemotherapy within the past 12 months
* Will attend a daycare facility that does not separate children by age and contains an infant who is less than 6 months of age during study days 0 to 28

Temporary Exclusion Criteria for RSV-Seropositive and RSV-Seronegative Children:

To be eligible to participate, RSV-seropositive and RSV-seronegative infants and children must satisfy none of the temporary exclusion criteria. The following conditions are temporary or self-limiting. Once the condition is resolved and the subject is otherwise eligible, the subject may be enrolled or rescreened, if necessary.

* Any of the following events at the time of inoculation:

  * fever (rectal temperature of greater than or equal to 100.4°F),
  * upper respiratory signs or symptoms (rhinorrhea, cough, or pharyngitis)
  * nasal congestion significant enough to interfere with successful inoculation
  * otitis media
* Receipt of any killed vaccine or live-attenuated rotavirus vaccine less than 14 days prior to inoculation
* Receipt of the following medications less than 28 days prior to inoculation:

  * any live vaccine other than rotavirus
  * another investigational vaccine or investigational drug,
  * systemic corticosteroids administered for greater than 14 days at a dosage equivalent to prednisone at greater than 2 mg/kg or 20 mg daily
  * salicylate (aspirin) or salicylate-containing products
* Receipt of a non-permitted concomitant medication or any of the following medications less than 3 days prior to inoculation:

  * systemic antibacterial, antiviral, antifungal, anti-parasitic, or antituberculous agents, whether for treatment or prophylaxis,
  * intranasal medications
* Scheduled administration of the following in relation to planned inoculation:

  * killed vaccine within the 14 days following,
  * any live vaccine other than rotavirus within the 28 days following,
  * another investigational vaccine or drug within the 28 days following for RSV-seropositive children and the 56 days following for RSV-seronegative infants and children

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-10; Primary Completion 2018-04-26 (Actual); Study Completion 2018-04-26 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related solicited adverse events (AEs) that occur during the acute monitoring phase of the study | Measured at days 0-10 for seropositive and days 0-28 for seronegative
Severity of vaccine-related solicited AEs that occur during the acute monitoring phase of the study | Measured at days 0-10 for seropositive and days 0-28 for seronegative
Frequency of vaccine-related lower respiratory illness | Measured during study days 0-28 for seropositive subjects and study days 0-56 for seronegative subjects
Proportion of subjects shedding vaccine virus | Measured during study days 0-28 for seropositive subjects and study days 0-56 for seronegative subjects
Proportion of subjects that develop 4-fold or greater increases in RSV neutralizing antibody titer following vaccination | Measured during study days 0-28 for seropositive subjects and study days 0-56 for seronegative subjects

CONTACTS AND LOCATIONS:
Overall Officials: Ruth A. Karron, MD, Principal Investigator — Center for Immunization Research (CIR), Johns Hopkins Bloomberg School of Public Health (JHSPH)
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

DOCUMENTS (1):
  • Informed Consent Form (2016-01-29): https://cdn.clinicaltrials.gov/large-docs/12/NCT02601612/ICF_000.pdf